CLINICAL TRIAL: NCT04516941
Title: Efficacy and Safety of Edoxaban and or Colchicine for Patients With SARS-CoV-2 Infection Managed in the Out of Hospital Setting
Brief Title: CorONa Virus edoxabaN ColchicinE (CONVINCE) COVID-19
Acronym: CONVINCE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient rate of patient accrual and newly available scientific evidence
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CONVINCE Version 1.0 12052020
Record Dates: First submitted 2020-08-05; First posted 2020-08-18 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV Infection; COVID-19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — edoxaban; Colchicine

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Edoxaban (Active Comparator): Edoxaban 60 mg q.d., or 30 mg q.d. in patients with CrCl = or <50 ml/min or body weight equal or less than 60 kg from randomization to end of study visit at day 25 (+/-3).
  Interventions: Drug: Edoxaban Tablets
- Colchicine (Active Comparator): Colchicine at 0.5 mg per os (PO) twice daily for the first 3 days and then once daily from randomization to day 14 (+/-3) days. Treatment could be continued to day 25 (+3/-3 days).
  Interventions: Drug: Colchicine Tablets
- No Edoxaban and No Colchicine (No Intervention): No intervention
- Edoxaban and Colchicine (Active Comparator): Edoxaban 60 mg q.d., or 30 mg q.d. in patients with CrCl = or <50 ml/min or body weight equal or less than 60 kg from randomization to end of study visit at day 25 (+/-3).
  Colchicine at 0.5 mg per os (PO) twice daily for the first 3 days and then once daily from randomization to day 14 (+/-3) days. Treatment could be continued to day 25 (+3/-3 days).
  Interventions: Drug: Edoxaban Tablets; Drug: Colchicine Tablets

INTERVENTIONS:
Drug: Edoxaban Tablets — Treatment
  Arms: Edoxaban; Edoxaban and Colchicine
Drug: Colchicine Tablets — Treatment
  Arms: Colchicine; Edoxaban and Colchicine

SUMMARY:
There is emerging evidence that patients with SARS-CoV-2 are affected by increased coagulopathy, including in the most advanced forms, a fully blown disseminated intravascular coagulation, leading to multi organ failure (MOF). Post-Morten observations from patients who died because of SARS-CoV-2 infection in Bergamo, Italy and other places have revealed the presence of diffuse venous, arterial and microcirculatorythrombosis, not only restricted to the lung but also involving the kidneys, heart and gut.

Thrombin plays a central role in mediating clot forming as well as in mediating inflammation. A direct factor X inhibitor, namely edoxaban can act as prophylactic measure to mitigate the risk of venous and arterial thrombotic complications.

Colchicine is an inexpensive (generic drug), orally administered, and a potent anti-inflammatory medication. It might accelerate SARS-CoV-2 clearance.

The aim of the CONVINCE study is therefore to assess the safety and efficacy of edoxaban and/or colchicine administration in SARS-CoV-2 infected patients who are managed outside the hospital with respect to the occurrence of fatalities, hospitalisation, major vascular thrombotic events or the SARS-CoV-2 clearance rate under RT PCR.

ELIGIBILITY:
Inclusion Criteria:

Patients with laboratory confirmed SARS-CoV-2 infection (under RT PCR) who are managed at home or in another out-of-hospital setting.

Exclusion Criteria:

Hepatic disease associated with coagulopathy and clinically relevant bleeding risk, including Child-Pugh C cirrhosis with portal hypertension.

* Lesion or condition, if considered to be a significant risk for major bleeding. This may include current or recent gastrointestinal ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial haemorrhage, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities.
* Uncontrolled severe hypertension.
* Ongoing or planned treatment with parenteral or oral anticoagulants
* Unilateral or bilateral above knee lower extremity amputation.
* Inability to take oral medication or otherwise unable or unwilling to undergo/perform study-specified procedures
* Have received or will receive an experimental drug or used an experimental medical device within 30 days before the planned start of treatment
* Pregnancy or breast-feeding or any plan to become pregnant during the study. Women (and men, for Colchicine group only) with child-bearing potential not using adequate birth control method (note: as adequate method of birth control oral contraception is recommended. If oral contraception is not feasible, both partners should use adequate barrier birth control).
* Need for dual anti-platelet therapy consisting of aspirin and an oral P2Y12 inhibitor
* Inflammatory bowel disease or chronic diarrhea or neuromuscular disease
* Creatinine clearance (CrCl) <15 ml/min
* Anticipated use of Hydroxychloroquine
* Participation in any other clinical trial
* Inability to understand the requirements of the study and to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Edoxaban vs. no active treatment | Baseline to day 25
  To assess the effect of edoxaban versus no active treatment on the composite endpoint of asymptomatic proximal deep-vein thrombosis, symptomatic proximal or distal deep-vein thrombosis, symptomatic pulmonary embolism or thrombosis, myocardial infarction, ischemic stroke, non-CNS systemic embolism or death at day 25 (+/-3) after randomization.
Colchicine vs no active treatment | Baseline to day 14
  To assess the effect of colchicine versus no active treatment on the SARS-CoV-2 clearance rates under RT PCR or freedom from death or hospitalisation at day 14 (+/-3) after randomization.

SECONDARY OUTCOMES:
Number of patients with asymptomatic proximal deep-vein thrombosis | Baseline to day 25
  An intraluminal filling defect on CT scan or MR venography in the IVC or iliac veins.
Number of patients with symptomatic proximal or distal deep-vein thrombosis | Baseline to day 25
  Typical symptoms of DVT associated with non-compressible vein segment on ultrasonography or an intra-luminal filling defect on venography, CT venography or MRI venography,located in the inferior vena cava (IVC), the iliac vein, the common femoral vein, the femoral or the popliteal vein.
Number of patient with symptomatic pulmonary embolism or thrombosis | Baseline to day 25
  Typical symptoms of PE associated with
  * an intra-luminal filling defect in (sub) segmental or more proximal branches on spiral computed tomography scan (CT) or computerized tomographic pulmonary angiography (CTPA).
  * a considerable perfusion defect (~ 75% of a segment) with a local normal ventilation result (high probability) during perfusion-ventilation lung scan (PLS, VLS or V/Q scan).
  * an intraluminal filling defect or a sudden cut-off of vessels (~more than 2.5 mm in diameter) on a catheter guided pulmonary angiogram.
  In case of an inconclusive CTPA, inconclusive V/Q scan or inconclusive angiography demonstration of DVT in the lower extremities e.g. by compression ultrasound or venography will be required
Number of patients with myocardial infarction | Baseline to day 25
  For the primary analysis, MI endpoint will be defined based on the third universal definition of myocardial infarction with the exception of periprocedural MI after PCI, which will be defined according to the SCAI definition.
Number of patients with ischemic stroke | Baseline to day 25
Number of patients with non-CNS systemic embolism | Baseline to day 25
  Ischemic stroke is defined as an acute episode of focal cerebral, spinal, or retinal dysfunction caused by CNS infarction
Number of deaths | Baseline to day 25
  Death will be classified in 5 categories with respect to cause. Thromboembolism, cardiovascular, bleeding, Pulmonary other known cause. In general, all deaths will be assumed to be due to thromboembolism or pulmonary in nature unless another cause is obvious
Ventilation need | Baseline to day 25
  Need for non-invasive or invasive ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, Prof. Dr., Study Chair — Bern University Hospital
Locations (5):
- Jessa Ziekenhuis, Hasselt, Belgium
- Italy (2):
  - ASST Rhodense, Garbagnate Milanese
  - ASST Grande Ospedal Metropolitano Niguardia, Milan
- Switzerland (2):
  - Ospedale regionale Lugano, Lugano, Canton Ticino
  - Bern University Hospital, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Result] Zhou F, Fan G, Liu Z, Cao B. SARS-CoV-2 shedding and infectivity - Authors' reply. Lancet. 2020 Apr 25;395(10233):1340. doi: 10.1016/S0140-6736(20)30869-2. Epub 2020 Apr 15. No abstract available. PMID 32304646
- [Result] Varga Z, Flammer AJ, Steiger P, Haberecker M, Andermatt R, Zinkernagel AS, Mehra MR, Schuepbach RA, Ruschitzka F, Moch H. Endothelial cell infection and endotheliitis in COVID-19. Lancet. 2020 May 2;395(10234):1417-1418. doi: 10.1016/S0140-6736(20)30937-5. Epub 2020 Apr 21. No abstract available. PMID 32325026
- [Result] Ranucci M, Ballotta A, Di Dedda U, Baryshnikova E, Dei Poli M, Resta M, Falco M, Albano G, Menicanti L. The procoagulant pattern of patients with COVID-19 acute respiratory distress syndrome. J Thromb Haemost. 2020 Jul;18(7):1747-1751. doi: 10.1111/jth.14854. Epub 2020 May 6. PMID 32302448
- [Result] Panigada M, Bottino N, Tagliabue P, Grasselli G, Novembrino C, Chantarangkul V, Pesenti A, Peyvandi F, Tripodi A. Hypercoagulability of COVID-19 patients in intensive care unit: A report of thromboelastography findings and other parameters of hemostasis. J Thromb Haemost. 2020 Jul;18(7):1738-1742. doi: 10.1111/jth.14850. Epub 2020 Jun 24. PMID 32302438
- [Result] Poissy J, Goutay J, Caplan M, Parmentier E, Duburcq T, Lassalle F, Jeanpierre E, Rauch A, Labreuche J, Susen S; Lille ICU Haemostasis COVID-19 Group. Pulmonary Embolism in Patients With COVID-19: Awareness of an Increased Prevalence. Circulation. 2020 Jul 14;142(2):184-186. doi: 10.1161/CIRCULATIONAHA.120.047430. Epub 2020 Apr 24. No abstract available. PMID 32330083
- [Derived] Landi A, Morici N, Vranckx P, Frigoli E, Bonacchini L, Omazzi B, Tresoldi M, Camponovo C, Moccetti T, Valgimigli M. Edoxaban and/or colchicine in outpatients with COVID-19: rationale and design of the CONVINCE trial. J Cardiovasc Med (Hagerstown). 2023 Dec 1;24(12):920-930. doi: 10.2459/JCM.0000000000001556. Epub 2023 Nov 3. PMID 37942793
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014